CLINICAL TRIAL: NCT04174625
Title: The Effect of Omega 3 Supplementations on Serum 25 Hydroxyvitamin D Levels
Brief Title: The Effect of Omega 3 on 25 Hydroxyvitamin D
Acronym: n-3FAon25OHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science Private University (Other)
Responsible Party: Principal Investigator, Mahmoud Suleiman Abu-Samak, Prof.Dr. Mahmoud Suleiman Abu-Samak, Applied Science Private University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DRGS-2014-2015-165-5
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: 25-hydroxyvitamin D Levels
Keywords: omega 3; 25 hydroxyvitamin D; 25OHD; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega3-FA group (Experimental): Omega3-FA group 1000 mg wild salmon and fish oil complex (contains 300 mg of omega3-FA) once daily
  Interventions: Dietary Supplement: Dietary Supplement: Omega3-FA
- Control group (Experimental): VD3 group 50,000 IU/week
  Interventions: Dietary Supplement: Dietary Supplement: Omega3-FA

INTERVENTIONS:
Dietary Supplement: Dietary Supplement: Omega3-FA — Dietary Supplement: Omega3-FA 300 mg of omega3-FA once daily for 8 weeks
  Other Names: n-3FA

SUMMARY:
The effect of omega 3 fatty acid on serum 25-hydroxyvitamin D levels.

DETAILED DESCRIPTION:
No data are available on the effect of omega 3 on serum 25-hydroxyvitamin D levels in Jordanian men and women.

This study was designed to investigate whether omega 3 supplementation has a potential effect on the reducing of serum 25-hydroxyvitamin D levels.

This randomized, placebo-controlled clinical trial (RCT) was designed to evaluate 300 mg omega-3FA daily for 2 months on serum levels of 25-hydroxyvitamin D levels. This RCT will be conducted on 80 to 90 Jordanian men and women aged 22 to 66 years. Baseline and follow-up levels for 25-hydroxyvitamin D (25OHD), parathyroid hormone (PTH), calcium, phosphate, liver and kidney functions will be assayed.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years old

Male and female Jordanian ASU students and employees who live in Amman.

Informed written consent from the participant prior to the start of the study.

a serum 25(OH)D concentration between 10 and 70 ng/mL.

Exclusion Criteria:

Any eligiable subject refuses to apply with informed written consent before the start of the study.

Men or women previously diagnosed with chronic diseases, including kidney disease or GIT problems.

Who are receiving vitamin D3 supplements (3 months before the start of the study) .

Pregnants,Breastfeeding females ,Females using hormonal contraceptives

Ages: 22 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2021-07-17 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
serum concentrations of 25-hydroxyvitamin D | 8 weeks
  ng/ml
serum concentrations of PTH | 8 weeks
  pg/mL

OTHER OUTCOMES:
serum concentration of calcium | 8 weeks
  mg/dl
serum concentration of phosphate | 8 weeks
  mg/dl
serum ALT | 8 weeks
  U/L
Serum urea | 8 weeks
  mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud S Abu-Samak, PhD, Principal Investigator — Department of Clinical Pharmacy and Therapeutics
Locations (1):
- Mahmoud S Abu-Samak, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: after six months
Access Criteria: open access